CLINICAL TRIAL: NCT07162324
Title: Prognostic Factors, Surgical Management and Survival of Glioblastoma Patients: a Multicenter Prospective Study
Brief Title: A Multicenter, Prospective Study for Glioblastoma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other); University of California, San Francisco (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Kostas N. Fountas, Professor & Chairman, Larissa University Hospital
Other Study IDs: 27446
Record Dates: First submitted 2025-08-06; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma
Keywords: glioblastoma; lobectomy; complications; outcome; overall survival; progression free survival
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Glioblastoma (GBM) is the most common and aggressive primary tumor of the adult central nervous system (CNS), with a poor prognosis and median overall survival ranging between 14 to 20 months despite advancements in diagnostic and therapeutic strategies. This prospective, observational, multicenter study aims to collect and analyze comprehensive data from GBM patients treated across selected centers in Europe and the United States, the investigators' centers included. Information will include demographics, imaging findings, molecular subtypes, clinical status, surgical strategies, postoperative management, complications, and follow-up data. Patients over 18 years old with radiographic evidence of GBM who provide informed consent will be included. Surgical interventions will vary, ranging from biopsy to supramaximal resections, based on individual patient and surgeon decisions. Key outcomes of interest include overall survival (OS) and progression-free survival (PFS). Secondary endpoints include perioperative complications, extent of resection (EoR), pre- and postoperative Karnofsky Performance Scores (KPS), hospital stay duration, and identification of risk factors influencing OS and functional outcomes. Patient monitoring will include standardized follow-up at one, three, and six months postoperatively, and quarterly thereafter or as clinically indicated. Statistical analysis will be conducted using R software, applying descriptive statistics, chi-square tests, logistic and linear regression, and assessing statistical significance at p < 0.05. Results will also be expressed in odds ratios with 95% confidence intervals. This study seeks to define optimal surgical strategies based on patient-specific factors and contribute to improved, personalized treatment pathways for GBM management.

DETAILED DESCRIPTION:
Brief Background: Glioblastoma remains the most prevalent and aggressive primary tumor of the Central Nervous system (CNS) in adults, with dismal prognosis and median overall survival between 14 to 20 months, despite the current advances in diagnostics and treatment options.

Aim: The aim of this study is to collect data prospectively in all glioblastoma patients treated in centers across Europe and the United States (US). In this data there will be included information regarding demographics, imaging, molecular subtypes, preoperative clinical status, surgical strategy in these patients, and post-operative management, along with any complications. Eventually this data will be assessed in order to distinguish the best surgical approach, according to different groups of patients (e.g. age, molecular subtype, tumor locations etc). Furthermore, treatment effect, tumor pseudo-progression, and recurrence management will also be assessed.

Study Design: This project constitutes a prospective, observational, multicenter study. The centers included are staffed with multiple experienced neurooncology surgeons. Patients will undergo a thorough demographic, family and medical history, and clinical examination. The patients' imaging studies will also be assessed. After the surgical management chosen, each patient will be closely monitored postoperatively until discharge. Postoperative imaging, postoperative neurological evaluation, and any complications will be thoroughly documented. Pathology reports, along with information regarding molecular subtypes will be included. The patients will be re-evaluated at one, three, and six months postoperatively, and then every three months or sooner in cases of any suspicion of recurrence or any changes in the patient's clinical status.

Patients: The investigators will include patients fulfilling the following eligibility criteria: Inclusion criteria:

* Adult patients (>18 years of age) with
* Glioblastoma based on radiographic features (Magnetic Resonance Imaging),
* Patients that consent for study participation.

Exclusion criteria:

* Non adult patients (<18 years of age),
* Patients that do not consent for participation in this study,
* Patients with other CNS tumors (primary or secondary). Intervention: Patients with tumors, compatible with glioblastomas -according to conventional Magnetic Resonance Imaging (MRI)- will fulfil their written consent and will then be included in the study. Each patient will be treated with a different surgical management (e.g biopsy, subtotal resection, gross-total resection, supramaximal resection or lobectomy) according to surgeons' and/or patients' choice. Any adjunct treatment will be documented (such as chemotherapy or/and radiotherapy).

Outcome: The primary endpoints of the study are: (1) The overall survival (OS) of the patients (2) The progression free survival (PFS) of the patients. OS and PFS will be calculated in months.

The secondary endpoints of the study are: (1) Peri- and post-operative complications, (2) Length of hospital stay counted in days, (3) Preoperative and postoperative Karnofsky Performance Scale (KPS) score (1-100), and (4) Extent of Resection (EoR) (counted as the % percentage of the preoperative tumor).

Co-registration of: (1) Risk factors affecting OS and PFS ( patient's age, cerebral dominance, BMI, tumor's molecular subtype),(2) Age (measured in years), (3) Gender (male, female, other), (4) Other demographic information (such as nationality, education level), (5) Anatomic location of the tumor, (6) Size of the tumor before intervention (measured in cm), (7) Intake of mannitol, hypertonic saline or steroids, (8) Dexterity, (9) Symptoms at the time of hospital admission, and (10) Molecular subtype of the tumor.

Timing: Follow up: one month, six months, and then every three months postoperatively. In cases of tumor recurrence or post-discharge complications patients will be reassessed. Enrollment of the first patient will take place after approval by the IRB and Research registration. Indicative time period: 2025 - 2030.

Statistical analysis: Descriptive statistics will be used to summarize count and continuous data. In particular, count data will be presented in absolute numbers and percentages, while continuous data will be given in mean (and standard deviation) or median values (and interquartile ranges) according to the Kolmogorov test. We will also use the chi-square test and logistic regression (or Kruskal-Wallis test), and linear regression to test for between-group differences. Statistical significance will be set at 0.05. All statistical analyses will be carried out in R statistical environment. For count data the results will also be provided in odds ratio along with their 95% confidence interval (CI).

ELIGIBILITY:
Inclusion criteria:

* Adult patients (>18 years of age) with
* Glioblastoma based on radiographic features,
* Patients that consent for study participation.

Exclusion criteria:

* Non adult patients,
* Patients that do not consent for participation in this study,
* Patients with other CNS tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioblastoma patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Five years
  Overall survival of glioblastoma patients will be measured in months
Progression Free Survival | Five years
  Progression Free Survival of glioblastoma patients will be measured in months.

SECONDARY OUTCOMES:
Peri- and postoperative complications | 3 months
  Peri- and postoperative complications
Length of hospital stay | 30 days
  Length of hospital stay, measured in days
Preoperative and post operative Karnofsky Performance Scale (KPS) score (1-100) | 5 years
  Preoperative and post operative Karnofsky Performance Scale (KPS) score (1-100)
Extent of Resection (EoR) | up to 48 hours
  Extent of Resection (EoR) (% percentage of the preoperative tumor)

CONTACTS AND LOCATIONS:
Overall Officials: Kostas Fountas, MD, PhD, Principal Investigator — University Hospital of Larisa,Greece; Mitchel Berger, MD, Study Director — Department of Neurosurgery, UCSF; Philippe Schucht, MD, PhD, Study Chair — University of Bern, Department of Neurosurgery
Locations (3):
- UCSF Weil Institute for Neurosciences, San Francisco, California, United States
- University Hospital of Larissa, Larissa, Thessaly, Greece
- Inselspital University Hospital of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arvaniti CK, Brotis AG, Young JS, Sivanrupan S, Menna G, Nishide M, Schucht P, Berger M, Fountas KN. The role of Lobectomy in Glioblastoma management: A Retrospective series. Brain Spine. 2025 Jun 18;5:104305. doi: 10.1016/j.bas.2025.104305. eCollection 2025. PMID 40678087
- [Background] Arvaniti CK, Karagianni MD, Papageorgakopoulou MA, Brotis AG, Tasiou A, Fountas KN. The Role of Lobectomy in Glioblastoma Management. Adv Tech Stand Neurosurg. 2025;55:137-151. doi: 10.1007/978-3-031-90762-3_7. PMID 40608104
- [Background] Arvaniti CK, Karagianni MD, Papageorgakopoulou MA, Brotis AG, Tasiou A, Fountas KN. The role of lobectomy in glioblastoma management: A systematic review and meta-analysis. Brain Spine. 2024 Apr 23;4:102823. doi: 10.1016/j.bas.2024.102823. eCollection 2024. PMID 39285857
- [Background] Louis DN, Perry A, Reifenberger G, von Deimling A, Figarella-Branger D, Cavenee WK, Ohgaki H, Wiestler OD, Kleihues P, Ellison DW. The 2016 World Health Organization Classification of Tumors of the Central Nervous System: a summary. Acta Neuropathol. 2016 Jun;131(6):803-20. doi: 10.1007/s00401-016-1545-1. Epub 2016 May 9. PMID 27157931
- [Background] Wach J, Vychopen M, Kuhnapfel A, Seidel C, Guresir E. A Systematic Review and Meta-Analysis of Supramarginal Resection versus Gross Total Resection in Glioblastoma: Can We Enhance Progression-Free Survival Time and Preserve Postoperative Safety? Cancers (Basel). 2023 Mar 15;15(6):1772. doi: 10.3390/cancers15061772. PMID 36980659
- [Background] Pessina F, Navarria P, Cozzi L, Ascolese AM, Simonelli M, Santoro A, Clerici E, Rossi M, Scorsetti M, Bello L. Maximize surgical resection beyond contrast-enhancing boundaries in newly diagnosed glioblastoma multiforme: is it useful and safe? A single institution retrospective experience. J Neurooncol. 2017 Oct;135(1):129-139. doi: 10.1007/s11060-017-2559-9. Epub 2017 Jul 8. PMID 28689368
- [Background] Eyupoglu IY, Hore N, Merkel A, Buslei R, Buchfelder M, Savaskan N. Supra-complete surgery via dual intraoperative visualization approach (DiVA) prolongs patient survival in glioblastoma. Oncotarget. 2016 May 3;7(18):25755-68. doi: 10.18632/oncotarget.8367. PMID 27036027
- [Background] Tripathi S, Vivas-Buitrago T, Domingo RA, Biase G, Brown D, Akinduro OO, Ramos-Fresnedo A, Sherman W, Gupta V, Middlebrooks EH, Sabsevitz DS, Porter AB, Uhm JH, Bendok BR, Parney I, Meyer FB, Chaichana KL, Swanson KR, Quinones-Hinojosa A. IDH-wild-type glioblastoma cell density and infiltration distribution influence on supramarginal resection and its impact on overall survival: a mathematical model. J Neurosurg. 2021 Oct 29;136(6):1567-1575. doi: 10.3171/2021.6.JNS21925. Print 2022 Jun 1. PMID 34715662
- [Background] De Bonis P, Anile C, Pompucci A, Fiorentino A, Balducci M, Chiesa S, Lauriola L, Maira G, Mangiola A. The influence of surgery on recurrence pattern of glioblastoma. Clin Neurol Neurosurg. 2013 Jan;115(1):37-43. doi: 10.1016/j.clineuro.2012.04.005. Epub 2012 Apr 24. PMID 22537870

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT07162324/Prot_SAP_000.pdf